CLINICAL TRIAL: NCT07394244
Title: Pucotenlimab Combined With Becotatug Vedotin in Advanced Cutaneous Squamous Cell Carcinoma: A Single-Arm, Multicenter, Prospective Phase II Clinical Trial
Brief Title: Pucotenlimab Combined With Becotatug Vedotin in Advanced Cutaneous Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Lepu Biopharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Deputy chief of medical oncology, chief physician，Fudan University Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Fudan CSCC-01
Record Dates: First submitted 2026-01-19; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cutaneous Squamous Cell Carcinoma (CSCC)
Keywords: Becotatug Vedotin; Pucotenlimab; CSCC; EGFR-ADC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Becotatug Vedotin+Pucotenlimab (Experimental): The medications are administered via intravenous infusion. Pucotenlimab is given at a fixed dose of 200 mg, and Becotatug Vedotin is dosed at 2.0 mg/kg based on the patient's actual body weight. The infusion time for each drug is 60 ± 15 minutes (if infusion-related reactions occur, the infusion duration may be extended, up to a maximum of 4 hours). Dosing occurs on the first day of each 3-week cycle (Q3W). Pucotenlimab and Vebreltus are administered on the same day, with Pucotenlimab given first. The infusion of Vebreltus should start at least 30 minutes after the completion of the Pucotenlimab infusion. For the first cycle, the infusion time for both drugs must not be less than 60 minutes.
  Interventions: Drug: Pucotenlimab; Drug: Becotatug Vedotin

INTERVENTIONS:
Drug: Pucotenlimab — The medications are administered via intravenous infusion. Pucotenlimab is given at a fixed dose of 200 mg, The infusion time is 60 ± 15 minutes (if infusion-related reactions occur, the infusion duration may be extended, up to a maximum of 4 hours). Dosing occurs on the first day of each 3-week cycle (Q3W). Pucotenlimab should be given first. For the first cycle, the infusion time for both drugs must not be less than 60 minutes.
  Other Names: HX008
Drug: Becotatug Vedotin — The medications are administered via intravenous infusion. Becotatug Vedotin is dosed at 2.0 mg/kg based on the patient's actual body weight. The infusion time for Becotatug Vedotin is 60 ± 15 minutes (if infusion-related reactions occur, the infusion duration may be extended, up to a maximum of 4 hours). Dosing occurs on the first day of each 3-week cycle (Q3W). The infusion of Becotatug Vedotin should start at least 30 minutes after the completion of the Pucotenlimab infusion. For the first cycle, the infusion time must not be less than 60 minutes.
  Other Names: MRG003

SUMMARY:
Study Design The study plans to enroll 38 patients. A Simon's two-stage design is employed. Based on historical data, the objective response rate (ORR) for patients meeting the inclusion criteria and receiving PD-1 inhibitor monotherapy is approximately 30%. The expected ORR for the combination of Pucotenlimab and Vebreltus is 55%. With a one-sided α=0.05 and 80% power, 9 patients will be enrolled in the first stage. If ≥2 patients achieve a partial response (PR) or complete response (CR), the study will proceed to the second stage. An additional 25 patients will be enrolled in the second stage, resulting in a total of 34 patients. If ≥15 patients in the total population achieve a PR, the study endpoint is considered met. Accounting for a 10% dropout rate, a total of 38 patients will be enrolled.

Study Procedures After providing full informed consent and passing screening, eligible subjects will receive treatment with Vebreltus 2.0 mg/kg and Pucotenlimab 200 mg. On the first day of each treatment cycle, patients will receive an intravenous infusion of Pucotenlimab (infusion duration: 60 min ± 15 min, with the first cycle infusion lasting no less than 60 minutes). At least 30 minutes after the completion of the Pucotenlimab infusion, the Vebreltus infusion will commence (infusion duration: 60 min ± 15 min, with the first cycle infusion lasting no less than 60 minutes). Patients will receive the combination therapy once every 3 weeks until completion of 2 years of treatment or until the occurrence of a protocol-defined treatment discontinuation event. Following the end of treatment, each subject will undergo a 30-day (+7 days) safety follow-up to monitor adverse events and clinically relevant events. Post-treatment survival follow-up will be conducted every 12 weeks (±7 days). For subjects who discontinue treatment for reasons other than disease progression/death and do not initiate new anti-cancer therapy, tumor imaging assessments will continue per the original schedule until disease progression, initiation of new anti-cancer therapy, withdrawal of consent, loss to follow-up, or death, whichever occurs first.

After enrollment, tumor response will be assessed according to RECIST v1.1 and iRECIST criteria. Imaging evaluations will be performed every 6 weeks (±7 days) from the first dose for the first 54 weeks, and then every 9 weeks (±7 days) thereafter (regardless of any delays in study drug administration), until iRECIST-confirmed progressive disease (iPD), initiation of new anti-cancer therapy, withdrawal of informed consent, loss to follow-up, or death, whichever occurs first.

Exploratory Analysis This study will analyze the correlation between biomarkers in patient tumor tissue/blood samples (e.g., EGFR expression, PD-L1 CPS score, TILs) collected before and after treatment and clinical efficacy endpoints (e.g., ORR, PFS, DoR).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and agree to comply with the protocol requirements.
2. Age ≥18 years and ≤80 years on the day of signing the informed consent form, regardless of gender.
3. Life expectancy ≥12 weeks.
4. Histopathologically confirmed cutaneous squamous cell carcinoma (cSCC), which is either locally advanced and inoperable (including recurrence after ≥2 prior surgeries, or deemed unresectable by a surgeon, or where surgery may lead to severe complications or deformity) or metastatic.
5. Have received 0-1 prior lines of systemic chemotherapy for advanced cSCC, and have experienced disease progression during or after the most recent treatment (relapse within 6 months after completing adjuvant therapy is considered as one line of therapy).
6. Able to provide tumor tissue specimens (paraffin blocks, paraffin-embedded sections, or fresh tissue sections) from a primary or metastatic site for pathological testing. The most recent archived tumor tissue specimen should be used. If archived tissue is unavailable, a new biopsy must be performed.
7. Have at least one measurable lesion at baseline according to RECIST 1.1 criteria (the longest diameter ≥10 mm on CT scan, or short axis ≥15 mm for lymph nodes; measurable lesions should not have been irradiated, unless progression has been demonstrated within a prior radiation field or after local therapy). Digital photography may be used for superficial lesions.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to treatment initiation.
9. No severe cardiac dysfunction, with left ventricular ejection fraction (LVEF) ≥50% within 28 days prior to treatment initiation.
10. Adequate organ function within 7 days prior to treatment initiation, defined as:

(1)Bone Marrow Function: Absolute neutrophil count (ANC) ≥1.5×10⁹/L, platelet count ≥100×10⁹/L, hemoglobin ≥90 g/L; and no transfusion or blood product administration within 14 days prior to the first dose, and no treatment with biologic response modifiers (e.g., G-CSF, erythropoietin) within 7 days prior to the first dose.

(2)Liver Function: For patients without liver metastases: total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN. For patients with liver metastases: TBIL ≤1.5 × ULN, ALT and AST ≤5 × ULN.

(3)Renal Function: Serum creatinine (Cr) ≤1.5 × ULN, or creatinine clearance (Ccr) ≥50 mL/min (calculated using the Cockcroft-Gault formula) (4)Coagulation Function: International normalized ratio (INR) ≤1.5 × ULN and activated partial thromboplastin time (APTT) ≤1.5 × ULN (unless the patient is receiving therapeutic anticoagulation).

11.Men and women of childbearing potential must agree to use effective contraception from the time of signing the informed consent form until 6 months after the last dose of the investigational product. Women of childbearing potential include premenopausal women and women within 2 years of menopause. A negative serum pregnancy test result is required for women of childbearing potential within ≤7 days before the first dose of the investigational product.

Exclusion Criteria:

1. History of other malignancies within the past five years, except for cured cervical carcinoma in situ, thyroid cancer, or cutaneous basal cell carcinoma.
2. Prior receipt of any of the following treatments:

   1. Any prior therapy targeting anti-PD-1, anti-PD-L1, PD-L2, CD137, CTLA-4 antibodies, or any other antibodies/drugs specifically targeting T-cell costimulation or immune checkpoint pathways;
   2. Any prior EGFR monoclonal antibody therapy;
   3. Investigational drug administration within 28 days before the first dose;
   4. Anticancer chemotherapy within 21 days before the first dose (washout period ≥14 days for oral fluoropyrimidines, leucovorin, or weekly paclitaxel chemotherapy; ≥42 days for nitrosoureas or mitomycin);
   5. Radiotherapy within 28 days before the first dose, or palliative radiotherapy for bone metastases within 2 weeks;
   6. Major surgery within 28 days before the first dose without full recovery, or planned major surgery within the first 12 weeks after receiving the study drug.
3. Symptomatic brain or leptomeningeal metastases (unless treated >6 months prior, with negative imaging within 4 weeks before enrollment, and stable neurological status without steroid therapy).
4. Any severe or uncontrolled systemic disease per investigator's judgment, including poorly controlled hypertension (systolic BP >160 mmHg or diastolic BP >100 mmHg), uncontrolled diabetes, or active bleeding signs.
5. Poorly controlled cardiac diseases, including NYHA Class II or higher heart failure, unstable angina, myocardial infarction within 1 year, or clinically significant supraventricular/ventricular arrhythmias requiring treatment.
6. Active infections, including:

   Hepatitis B (HBsAg-positive AND HBV DNA ≥2000 IU/mL, excluding drug-induced or other non-viral hepatitis);

   Hepatitis C (anti-HCV antibody-positive AND HCV RNA above the lower limit of detection);

   HIV infection; or uncontrolled active bacterial, viral, fungal, rickettsial, or parasitic infections (unless treated and resolved before study drug initiation).
7. History of hypersensitivity to any component of Pucotenlimab or Vebreltus (e.g., histidine, histidine hydrochloride, sucrose, mannitol, polysorbate 80), or ≥Grade 3 allergic reactions to macromolecular protein preparations/monoclonal antibodies.
8. Primary immunodeficiency history or active autoimmune disease requiring immunosuppressants or systemic glucocorticoids (dose ≥10 mg/day prednisone or equivalent within 2 weeks before enrollment).

   Note: Patients with type I diabetes, stable hypothyroidism on hormone replacement, psoriasis/eczema not requiring systemic therapy, or vitiligo may be enrolled. Topical/inhaled corticosteroids or short-term (≤7 days) glucocorticoid use for non-autoimmune conditions are exempted.
9. History or presence of interstitial lung disease, radiation pneumonitis, severe chronic obstructive pulmonary disease, severe respiratory insufficiency, or symptomatic bronchospasm.
10. Positive serum pregnancy test, lactation, or unwillingness to use adequate contraception during the study and for 6 months after the last dose.
11. Other conditions deemed inappropriate for participation by the investigator (e.g., alcohol/drug abuse).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-09 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 2 years
  ORR is defined as the proportion of subjects achieving confirmed Complete Response (CR) or Partial Response (PR) as assessed by the investigator according to RECIST v1.1 and iRECIST criteria. ORR analysis will be based on the Full Analysis Set (FAS)

SECONDARY OUTCOMES:
Disease Control Rate | up to 2 years
  Disease Control Rate (DCR) is defined as the proportion of subjects assessed by the Independent Review Committee (IRC) according to RECIST v1.1 criteria who achieve CR, PR, or Stable Disease (SD) (lasting for at least 6 weeks from the first dose), along with the exact 95% CI using the Clopper-Pearson method.
Progression-Free Survival | up to 2 years
  Progression-Free Survival (PFS) is defined as the time from enrollment to the first occurrence of disease progression or death from any cause. For subjects without observed progression or death, PFS will be censored at the time of the last valid and adequate assessment. PFS analysis will be based on the FAS. The median PFS and its 95% CI will be estimated using the Kaplan-Meier method, and progression-free survival curves will be generated.
Duration of Response | up to 2 years
  Duration of Response (DOR) is defined as the time from the first documented evidence of response (PR or CR according to RECIST v1.1 and iRECIST criteria, whichever is later) to the first documented disease progression (PD) or death from any cause, whichever occurs first, in subjects with a confirmed response. For subjects without observed progression or death, DOR will be censored at the time of the last adequate tumor assessment. DOR analysis will be performed on subjects who achieve CR or PR. The median DOR and its 95% CI will be estimated using the Kaplan-Meier method, and duration of response curves will be generated.
Overall Survival | up to 2 years
  Overall Survival (OS) is defined as the time from enrollment to death from any cause. For subjects not followed up to death, OS will be censored at the time of the last valid survival follow-up. Based on the FAS, the median OS (if applicable) and its 95% CI will be estimated using the Kaplan-Meier method, and survival curves will be plotted.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cencer Center, Shanghai, Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: No